CLINICAL TRIAL: NCT03105024
Title: Enhancing Exposure: the Impact of Self-efficacy Enhancement on Treatment Outcome
Brief Title: Self-efficacy Enhancement and Exposure Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Armin Zlomuzica, Dr. / Principal Investigator, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FP 1-1
Record Dates: First submitted 2017-03-27; First posted 2017-04-07 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Specific Phobia
Keywords: specific phobia; height phobia; exposure; virtual reality; extinction; self-efficacy
MeSH Terms: conditions — Phobia, Specific

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exposure + self-efficacy enhancement (Experimental): After the virtual exposure session, participants will receive instructions to recall the exposure session with a focus on the personal mastery experiences/achievements made during exposure.
  Interventions: Other: Self-efficacy enhancement
- Exposure + control intervention (Active Comparator): After the virtual exposure session, participants will receive instructions to recall the exposure session
  Interventions: Other: Control intervention
- Exposure only (No Intervention): Treatment as usual: no intervention after the exposure session will be given.

INTERVENTIONS:
Other: Self-efficacy enhancement — specific instructions regarding the retrieval of mastery experiences during exposure will be given (e.g., pointing out discrepancies between expected negative consequences and actual outcome during exposure; focus on achievements)
  Arms: Exposure + self-efficacy enhancement
Other: Control intervention — specific instructions regarding the retrieval of the exposure session will be given without an emphasis on personal mastery experience (e.g., description of details regarding the virtual reality environment)
  Arms: Exposure + control intervention

SUMMARY:
Self-efficacy refers to the perceived belief to cope effectively, by personal efforts, with challenging situations and problems (Bandura, 1977). Basic research has shown that increases in perceived self-efficacy can enhance the extinction of fear (Zlomuzica et al., 2015). This study is aimed at translating these findings into a useful clinical application to augment exposure-based treatment outcome.

DETAILED DESCRIPTION:
In this study, the effects of self-efficacy enhancement on treatment outcome in patients with height phobia will be investigated.

Participants will be randomly assigned to one of the following conditions: i) virtual reality exposure + self-efficacy enhancement; ii) virtual reality exposure + control intervention; iii) virtual reality exposure only. The amount of exposure is identical across groups (i.e. maximum of 1 hour of exposure). The self-efficacy and the control intervention involve the retrieval of the exposure session with or without a focus on personal mastery experiences/achievements, respectively.

Treatment-induced changes as well as the effects of self-efficacy enhancement will be measured on the subjective level (i.e. in-vivo Behavioral Approach Tests, BATs; church tower), physiological level (heart rate during the BATs), and subjective level (subjective fear during the BATs as well as height-phobia related questionnaires) at each of the three assessments (i.e. pretreatment, after which the exposure will conducted on the same day, i.e. day 1; posttreatment, which is scheduled approximately 2-3 days after exposure, and follow-up assessment, which will take place 1-month after exposure).

ELIGIBILITY:
Inclusion Criteria:

* specific phobia (acrophobia)
* normal or corrected vision

Exclusion Criteria:

* somatic or neurological disease
* personality disorder
* bipolar disorder
* acute drug- or alcoholabuse
* pharmacological treatment within the past 4 weeks
* mental retardation
* any schizophrenic disease

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
Change in the Behavioral Approach Test (BAT) | from pretreatment through follow-up (i.e. baseline, approx. 2-3 days after treatment, 1 month after)
Change in subjective fear during the BAT | from pretreatment through follow-up (i.e. baseline, approx. 2-3 days after, 1 month after)
  Subjective fear during the BATs will be measured using the Subjective Units of Distress Scale (SUDS)
Change in heart rate reactivity during the BAT | from pretreatment through follow-up (i.e. baseline, approx. 2-3 days after, 1 month after)

SECONDARY OUTCOMES:
Change in Acrophobia Questionnaire (AQ) | assessed from pre-treatment through follow-up (i.e. baseline, approx. 2-3 days after, 1 month after
Change in Attitude Towards Heights Questionnaire (ATHQ) | assessed from pre-treatment through follow-up (i.e. baseline, approx. 2-3 days after, 1 month after
Change in Danger Expectancy Scale (DES) | assessed from pre-treatment through follow-up (i.e. baseline, approx. 2-3 days after, 1 month after
Change in Anxiety Expectancy Scale (AES) | assessed from pre-treatment through follow-up (i.e. baseline, approx. 2-3 days after, 1 month after

OTHER OUTCOMES:
Change in perceived self-efficacy | assessed three times on day 1: before and after the exposure session as well as after the intervention; assessed once at posttreatment (window: 2-3 days after exposure treatment); assessed once at follow-up (window: 1 month after treatment)
  Changes in perceived self-efficacy will be measures with visual analogue scales (VAS)
Becks Depression Inventory II (BDI II) | assessed at pre-treatment (day 1)
State-Trait Anxiety Inventory (STAI) | assessed at pre-treatment (day 1)
Emotion Regulation Questionnaire (ERQ) | assessed at pre-treatment (day 1)
General Self-efficacy Scale (GSE) | assessed at pre-treatment (day 1)
Self-efficacy Scale (SES) | assessed at pre-treatment (day 1)
Resilience Appraisal Scale (RAS) | assessed after the intervention on day 1
Salivary cortisol | assessed twice at each of the three assessments, i.e. pretreatment, posttreatment, follow-up (windows: pretreatment on day 1; approx. 2-3 days after; 1 month after)
Changes in "Test zum kognitiven Schätzen" (TKS) | assessed twice on day 1: before and after exposure treatment

CONTACTS AND LOCATIONS:
Overall Officials: Armin Zlomuzica, Dr., Principal Investigator — Ruhr-University Bochum
Locations (1):
- Mental Health Research and Treatment Center, Bochum, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zlomuzica A, Preusser F, Schneider S, Margraf J. Increased perceived self-efficacy facilitates the extinction of fear in healthy participants. Front Behav Neurosci. 2015 Oct 16;9:270. doi: 10.3389/fnbeh.2015.00270. eCollection 2015. PMID 26528152
- [Background] Bandura A. Self-efficacy: toward a unifying theory of behavioral change. Psychol Rev. 1977 Mar;84(2):191-215. doi: 10.1037//0033-295x.84.2.191. No abstract available. PMID 847061